CLINICAL TRIAL: NCT06522724
Title: The Impact of Education on the Rehabilitation of Patients Hospitalized Due to Pneumonia With Confirmed COVID-19
Brief Title: Education Impact on Rehabilitation of Hospitalized Patients With Pneumonia and COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Renata Borys, MSc, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URzeszow 1/07/2021
Record Dates: First submitted 2024-07-19; First posted 2024-07-26 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Pneumonia Due to COVID-19
Keywords: pulmonary rehabilitation; COVID-19; pneumonia; patients' education
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: random selection to two groups (study group and control group)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education program and Pulmonary rehabilitation (Experimental): Conventional pulmonary rehabilitation coupled with original education program.
  Interventions: Other: Education program; Other: Pulmonary rehabilitation
- Pulmonary rehabilitation (Other): Conventional pulmonary rehabilitation
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Education program — Patients in a study group will participate in daily education program using an original brochure containing information about self-management during the treatment process, the benefits of appropriately adapted physical activity, practical tips on airway clearance techniques or physical exercise.
  Arms: Education program and Pulmonary rehabilitation
Other: Pulmonary rehabilitation — The patients will participate in a 14-day rehabilitation program (Monday to Saturday). Treatments and therapies will be continued for a maximum of three hours daily. The program will be applied individually to each patient and include in-bed assisted exercises, airway clearance techniques, effective cough exercises, pursed-lips breathing, exercises to strengthen the diaphragm and intercostal muscles and cardiopulmonary exercises.

SUMMARY:
The planned research will enable the assessment of rehabilitation's effects using two pulmonary rehabilitation models: conventional and supplemented with an education program for patients hospitalized due to pneumonia with confirmed COVID-19.

DETAILED DESCRIPTION:
The planned group size is 60 patients diagnosed with pneumonia and confirmed COVID-19. The given population was calculated based on the sampling calculator, considering the following parameters: fraction size, confidence level, and maximum error. Eligible patients will be randomly divided into two groups: a study group (30 patients) undergoing pulmonary rehabilitation supplemented with an education program, and a control group (30 patients) undergoing conventional pulmonary rehabilitation. Patients of both groups will be included in a 14-day rehabilitation program (Monday to Saturday). Treatments and therapies will be continued for a maximum of three hours daily. The program will be applied individually to each patient and include in-bed assisted exercises, airway clearance techniques, effective cough exercises, pursed-lips breathing, exercises to strengthen the diaphragm and intercostal muscles and cardiopulmonary exercises. Patients from the study group will additionally undergo daily education using an original brochure containing information about self management during the treatment process, the benefits of appropriately adapted physical activity, practical tips on airway clearance techniques or physical exercise. The test will be performed two times: before the start of rehabilitation and after completing the rehabilitation program. The patients' condition and the rehabilitation effects will be assessed using the following measures:

* Vital capacity (Voldyne 5000)
* Oxygen saturation (pulse oximeter)
* Acid-base balance (gasometry)
* Fatigue (modified Borg scale)
* Physical performance (Sit-to-Stand Test)
* Dyspnea assessment (MRC dyspnea scale)
* Anxiety and depression (HADS scale)
* Activities of daily living (Barthel scale)

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization due to pneumonia due to COVID-19
* Positive SARS-COV-2 PCR test
* Independence in in-bed sitting position with lower extremities placed on the floor
* Age 40 y.o. to 70 y.o.
* No additional respiratory support (e.a. cardiopulmonary bypass machine, ventilator)
* Informed, voluntary consent to participate in research.

Exclusion Criteria:

* Hospitalization due to pneumonia with negative SARS-COV-2 PCR test
* Unstable medical condition hindering performing the examination
* Age under 40 y.o. and over 70 y.o.
* Cognitive deficits impairing the ability to understand and execute commands
* Concomitant oncological, neurological, orthopedic, and psychiatric diseases may affect the examined persons' circulatory and respiratory functions, functional efficiency, quality of life, and emotional state.
* Failure to complete a 14-day rehabilitation program
* Lack of informed, voluntary consent to participate in research

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-10-26 (Actual)

PRIMARY OUTCOMES:
Vital capacity (Voldyne 5000) | First examination- before the start of the 14-day rehabilitation program
  Measurements will be performed with certified motivational spirometer, Voldyne 5000. Patient, in a sitting position, will inhale as much air as possible starting from residual volume (RV) level and approach to vital capacity (VC) level. The result will be read from the scale placed on the wall of the device.
Vital capacity (Voldyne 5000) | Second examination- at the end of the 14-day rehabilitation program
  Measurements will be performed with certified motivational spirometer, Voldyne 5000. Patient, in a sitting position, will inhale as much air as possible starting from residual volume (RV) level and approach to vital capacity (VC) level. The result will be read from the scale placed on the wall of the device.
Oxygen saturation | First examination- before the start of the 14-day rehabilitation program
  Measurements will be performed with pulse oximeter and the parameter analyzed will be SpO2 (oxygen saturation by pulse oximetry; percentage of oxygen in patients' blood).
Oxygen saturation | Second examination- at the end of the 14-day rehabilitation program
  Measurements will be performed with pulse oximeter and the parameter analyzed will be SpO2 (oxygen saturation by pulse oximetry; percentage of oxygen in patients' blood).
Acid-base balance | First examination- before the start of the 14-day rehabilitation program
  The gasometry results will be taken from patients' medical documentation. The parameters analyzed will be oxygen pressure (pO2) and carbon dioxide pressure (pCO2).
Acid-base balance | Second examination- at the end of the 14-day rehabilitation program
  The gasometry results will be taken from patients' medical documentation. The parameters analyzed will be oxygen pressure (pO2) and carbon dioxide pressure (pCO2).

SECONDARY OUTCOMES:
Physical performance assessment by Sit-to-Stand Test (STS) | First examination- before the start of the 14-day rehabilitation program
  The test will be performed starting in sitting position in the chair with straight back, feet flat on the floor, and arms crossed over the chest or placed on the thighs. The patient will be instructed to stand up fully from the seated position and then sit back down as quickly and safely as possible during 30 seconds (number of standings in 30 seconds).
Physical performance assessment by Sit-to-Stand Test (STS) | Second examination- at the end of the 14-day rehabilitation program
  The test will be performed starting in sitting position in the chair with straight back, feet flat on the floor, and arms crossed over the chest or placed on the thighs. The patient will be instructed to stand up fully from the seated position and then sit back down as quickly and safely as possible during 30 seconds (number of standings in 30 seconds).
Fatigue assessment using modified Borg scale | First examination- before the start of the 14-day rehabilitation program
  Fatigue will be examined during physical activity and the level of fatigue will be marked on a scale from 1 (no fatigue) to 10 (very very hard fatigue).
Fatigue assessment using modified Borg scale | Second examination- at the end of the 14-day rehabilitation program
  Fatigue will be examined during physical activity and the level of fatigue will be marked on a scale from 1 (no fatigue) to 10 (very very hard fatigue).
Dyspnea assessment with Medical Research Council dyspnea scale | First examination- before the start of the 14-day rehabilitation program
  Perceived breathlessness degree will be marked on a scale 0 (no breathlessness) to 4 (breathlessness at rest).
Dyspnea assessment with Medical Research Council dyspnea scale | Second examination- at the end of the 14-day rehabilitation program
  Perceived breathlessness degree will be marked on a scale 0 (no breathlessness) to 4 (breathlessness at rest).
Anxiety and depression assessment using HADS scale | First examination- before the start of the 14-day rehabilitation program
  The scale consists of 16 statements to which the respondent refers on a four-point scale. Eight statements are used to measure anxiety and depression, each of which is rated on a scale of 0 to 3 points. The cut-off threshold is 7 points for depression and 7 points for anxiety. The intensity of depressed mood and anxiety will be analyzed.
Anxiety and depression assessment using HADS scale | Second examination- at the end of the 14-day rehabilitation program
  The scale consists of 16 statements to which the respondent refers on a four-point scale. Eight statements are used to measure anxiety and depression, each of which is rated on a scale of 0 to 3 points. The cut-off threshold is 7 points for depression and 7 points for anxiety. The intensity of depressed mood and anxiety will be analyzed.
Activities of daily living assesment using Barthel scale | First examination- before the start of the 14-day rehabilitation program
  The Barthel Scale will be used to measure patient's ability to perform activities of daily living (ADLs) independently, with scores ranging from 0 (completely dependent) to 100 (completely independent).
Activities of daily living assesment using Barthel scale | Second examination- at the end of the 14-day rehabilitation program
  The Barthel Scale will be used to measure patient's ability to perform activities of daily living (ADLs) independently, with scores ranging from 0 (completely dependent) to 100 (completely independent).

CONTACTS AND LOCATIONS:
Overall Officials: Renata Borys, MSc, Principal Investigator — University of Rzeszow; Agnieszka Guzik, A/Prof, Study Director — University of Rzeszow; Magdalena Kołodziej, PhD, Study Chair — University of Rzeszow
Locations (1):
- University of Rzeszów, Rzeszów, Poland